CLINICAL TRIAL: NCT03494452
Title: Trunk Muscle Strength, Strength Endurance and Activity in Persons With Low Back Pain
Acronym: TRUSC
Status: Completed | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Other Study IDs: 2017-01714
Record Dates: First submitted 2018-02-27; First posted 2018-04-11 (Actual); Last update posted 2019-09-30 (Actual); Status verified 2019-09

CONDITIONS: Low Back Pain
Keywords: electromyography, strength, strength endurance
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Low back pain - no intervention: Patients who perform sitting occupational activities for at least 4 hours/day and have had low back pain for at least the previous 6 months
  Interventions: Other: No intervention
- Healthy - no intervention: Healthy persons who perform sitting occupational activities for at least 4 hours/day
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — There is no intervention in this cross-sectional study

SUMMARY:
The research questions are if persons with low back pain (LBP) have lower trunk muscle strength, lower trunk muscle strength endurance and lower trunk muscle activity than healthy controls and if functional limitations because of LBP are related to the level of muscle strength, strength endurance and activity. To investigate this investigators will carry out a clinical assessment including questionnaires and a biomechanical assessment comprising muscle strength tests, muscle strength endurance tests and electromyographic (EMG) analysis of selected trunk muscles.

DETAILED DESCRIPTION:
Objectives

The current state of research in the field and of the investigators own clinical experience clearly shows that the role of trunk muscle function in LBP is poorly understood. Investigators will address the following research questions:

* Do persons with LBP have lower trunk muscle strength, lower trunk muscle strength endurance and lower trunk muscle activity than healthy controls?
* Are functional limitations because of LBP related to the level of muscle strength, strength endurance and activity?

To answer these questions, investigators will establish an experimental framework to study limitations in muscle function to address the following aims:

* To compare trunk muscle strength, strength endurance and activity between persons with LBP and healthy control persons.
* To determine the relationship between trunk muscle strength, strength endurance and activity, and the Oswestry Disability Index (ODI) score.

The experimental setting consists of a clinical assessment using a questionnaire and a biomechanical assessment comprising muscle strength tests, muscle strength endurance tests and electromyographic analysis. Electromyographic activity of selected trunk muscles will be recorded during isokinetic and isometric trunk flexion and extension strength tests and during isometric trunk flexion and extension strength endurance tests.

Hypotheses Investigators hypotheses are that i. persons with LBP have lower trunk muscle strength, strength endurance and activity than healthy controls subjects. ii. the intensity of the EMG signal in lower back muscles decreases faster during the strength endurance test in persons with LBP than in healthy control subjects. iii. clinical scores correlate with trunk muscle strength, strength endurance and activity.

Procedures First, written informed consent will be obtained before participants will undergo a clinical exam (inspection and palpation of the lower back, measurement of active range of motion) performed by a trained physical therapist (PS). All participants will complete questionnaires to obtain pain and functional scores and information on their typical physical activity level (approximate duration: 30 minutes). Bipolar skin electrodes will be placed on selected trunk muscles (approximate duration: 15 minutes) and participants will walk on a treadmill for 10 min (warm-up). Participants will be seated on a strength testing system and practice trunk flexion and extension movements for 1 min. Subsequently, subjects will be asked to perform isokinetic trunk flexion and extension tests at maximum effort. EMG signals of the trunk muscles will be recorded during the maximum isokinetic contractions (approximate duration: 20 minutes). Subsequently, subjects will lie supine on a bench with their legs and pelvis supported by the bench. Their upper legs will be secured to the bench using a 15 cm wide Velcro belt. Subjects will be asked to hold their trunk in a horizontal position as long as possible while EMG signals of the trunk muscles will be recorded (approximate duration: 5 minutes).

ELIGIBILITY:
Inclusion Criteria:

* age ≥ 20 years
* age ≤ 55 years
* primarily seated occupational activities for at least 4 hours per working day
* patients:
* low back pain for at least 12 weeks

Exclusion Criteria:

* neurological symptoms
* diagnosed spinal damage
* cancer,or infectious diseases that could lead to chronic LBP
* other diseases that could affect physical performance
* surgery for chronic LBP
* pregnancy

Ages: 20 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: 20 persons with LBP 20 age and sex matched healthy control persons
Sampling Method: Non-Probability Sample
Enrollment: 36 (Actual)
Dates: Start 2017-10-10 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2019-05-31 (Actual)

PRIMARY OUTCOMES:
Isokinetic trunk muscle flexion strength | 0 months
  Maximum moment of isokinetic movement performed on a Biodex
Isokinetic trunk muscle extension strength | 0 months
  Maximum moment of isokinetic movement performed on a Biodex

SECONDARY OUTCOMES:
Trunk muscle activity | 0 months
  The rate of change in frequency and intensity of the EMG signal during the strength endurance test for the Mm. rectus abdominis, obliquus internus, obliquus externus, erector spinae longissimus, erector spinae iliocostalis, multifidus muscles
Isometric trunk muscle strength endurance | 0 months
  Biering-Soerensen test completion time of the will be recorded when the upper part of the body descended below the horizontal line
Back pain | 0 months
  visual analogue scale ranging from 0 (= no pain) to 10 (= worst pain)
Range of motion lumbar spine | 0 months
  Range of motion lumbar spine using the Schober test
Typical physical activity | 0 months
  Typical physical activity will be assessed using the self-administered short version of the German version of the International Physical Activity Questionnaire (IPAQ)
Disability | 0 months
  Disability will be assessed using the Oswestry Disability Index (ODI)

CONTACTS AND LOCATIONS:
Overall Officials: Annegret Muendermann, PhD, Principal Investigator — University Hospital, Basel, Switzerland
Locations (1):
- University Hospital Basel, Basel, Canton of Basel-City, Switzerland

IPD SHARING:
Plan to Share IPD: No